CLINICAL TRIAL: NCT01109108
Title: Streptococcus Pneumonia: Herd Effects and Emergence of Potentially Virulent Serotypes PCV13_Impact of NP Colonization, Herd Effects and Emergence of Potentially Virulent Serotypes of Pneumococci
Brief Title: Streptococcus Pneumonia: Effects of PCV13 on Pneumococcal Carriage
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Stephen Pelton, Professor of Pediatrics and Epidemiology, Boston Medical Center
Other Study IDs: H-28757
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-01

CONDITIONS: Nasopharyngeal Carriage of S. Pneumoniae
Keywords: pneumococcal vaccine; nasopharyngeal carriage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — NP specimens and bacterial isolates of S. pneuomoniae and nontypable Haemophilus
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children <2 years of age: Children <2 years of age with and without respiratory tract infection
- Children 2<5 years of age: Children 2<5 years of age with and without respiratory tract infection

SUMMARY:
The specific aim is to evaluate the impact of PCV13 as administered in the pediatric primary care clinic at Boston medical center on the serotype specific carriage of Streptococcus pneumoniae in children < 5.

Specifically the investigators will measure the decline in vaccine serotypes, the proportion of children receiving vaccine required to achieve 50% reduction in serotype specific carriage and the correlation between immunogenicity of the specific serotypes and decline in carriage. The study has been extended to complete 5 years of surveillance to determine the new SP serotype distribution at the time presumably a new equilibrium has been achieved.

ELIGIBILITY:
Inclusion Criteria:

* children < 5 years of age receiving care at Primary Care center at BMC and as many parent(s) as willing to participate

Exclusion Criteria:

* children with facial malformations making NP sampling unacceptable
* children in foster care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: children < 5 years of age receiving care at Primary Care center at BMC and as many parent(s) as willing to particpate
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2010-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Primary Care, Boston Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children aged 0<60 months with non-toxic appearance presenting for well child or urgent care visit at urban hospital recruited from July 1, 2010 - March 27, 2015; each child could be enrolled only once per 60 day period.
Groups:
- Children 0<2 Years of Age: Children 0<2 years of age with and without respiratory tract infection
Period: Overall Study
Arm/Group | Children 0<2 Years of Age | Children 2<5 Years of Age
Started | 4035 | 4755
Completed | 4035 | 4755
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Children 0<2 Years of Age: Children 0<2 years of age with and without concurrent respiratory tract infection
- Children 2<5 Years of Age: Children 2<5 years of age with and without concurrent respiratory tract infection
- Total: Total of all reporting groups
Arm/Group | Children 0<2 Years of Age | Children 2<5 Years of Age | Total
Number analyzed (Participants) | 4035 | 4755 | 8790
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4035 | 4755 | 8790
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 12.1 (5.7) | 40.0 (10.3) | 27.2 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1935 | 2402 | 4337
  Male | 2100 | 2353 | 4453
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 6 | 13
  Asian | 123 | 124 | 247
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2719 | 3445 | 6164
  White | 445 | 351 | 796
  More than one race | 739 | 828 | 1567
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4035 | 4755 | 8790
Pneumococcal risk factors [Count of Participants; unit: Participants]
  Current RTI (Respiratory tract infection): Yes | 1839 | 2108 | 3947
  Current RTI (Respiratory tract infection): No | 2196 | 2647 | 4843
  Recent antibiotic use (last 14 days): Yes | 535 | 451 | 986
  Recent antibiotic use (last 14 days): No | 3500 | 4304 | 7804
  Ever Breastfed: Yes | 3222 | 3684 | 6906
  Ever Breastfed: No | 813 | 1071 | 1884
  Current daycare attendance: Yes | 1217 | 2887 | 4104
  Current daycare attendance: No | 2818 | 1868 | 4686
  PCV13 Immune: Yes | 3240 | 3923 | 7163
  PCV13 Immune: No | 795 | 832 | 1627

OUTCOME MEASURES:

1. Primary Outcome: Nasopharngeal Colonization With PCV13 S. Pneumoniae
Description: Proportion of PCV13 serotypes among n=1851 children colonized with any S. pneumoniae
Time Frame: Study years 1-5
Population: Children colonized with any S. pneumoniae (PCV and non-PCV serotypes)
Measure: Count of Participants; unit: Participants
Arm/Group | Children 0<2 Years of Age | Children 2<5 Years of Age
Number analyzed (Participants) | 882 | 969
Participants
  2010-2011: number analyzed (Participants) | 186 | 168
  2010-2011: PCV13 serotype | 20 | 31
  2010-2011: Non-PCV13 serotype | 166 | 137
  2011-2012: number analyzed (Participants) | 329 | 308
  2011-2012: PCV13 serotype | 23 | 11
  2011-2012: Non-PCV13 serotype | 306 | 297
  2012-2013: number analyzed (Participants) | 193 | 244
  2012-2013: PCV13 serotype | 6 | 5
  2012-2013: Non-PCV13 serotype | 187 | 239
  2013-2014: number analyzed (Participants) | 110 | 155
  2013-2014: PCV13 serotype | 2 | 5
  2013-2014: Non-PCV13 serotype | 108 | 150
  2014-2015: number analyzed (Participants) | 64 | 94
  2014-2015: PCV13 serotype | 0 | 2
  2014-2015: Non-PCV13 serotype | 64 | 92
Statistical Analysis 1: Comparison: Children 2<5 Years of Age; Test type: Other; p < 0.05, Chi-squared; Risk Ratio (RR) = 1.0

ADVERSE EVENTS:
Arm/Group | Children <2 Years of Age | Children 2<5 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/4035 | 0/4755
Serious Adverse Events (participants affected / at risk) | 0/4035 | 0/4755
Other Adverse Events (participants affected / at risk) | 0/4035 | 0/4755

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes